CLINICAL TRIAL: NCT03378401
Title: Randomized, Placebo-controlled, Parallel Group, Double-blind, Multi-center Phase III Study to Assess the Inhibition of Plaque Formation of 0.1% Octenidine Mouthwash vs Placebo in Subjects With a Gingival Index ≤1.5
Brief Title: Study to Assess the Inhibition of Plaque Formation in Subjects With a Gingival Index ≤1.5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Schülke & Mayr GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OML-III-B; 2017-001698-18 (EudraCT Number)
Record Dates: First submitted 2017-12-11; First posted 2017-12-19 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Inhibition of Plaque Formation (by Gingivitis-Index ≤1.5)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Octenidine Mouthwash (Experimental): 0.1% Octenidinedihydrochlorid Solution for oromucosal use, mouth rinse with 10 ml for 30 s, 10 applications over 5 days
  Interventions: Drug: Octenidinedihydrochlorid
- Placebo (Placebo Comparator): Placebo Solution for oromucosal use, mouth rinse with 10 ml for 30 s, 10 applications over 5 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Octenidinedihydrochlorid — Mouth rinsing of the oral cavity with Octenidinehydrochlorid vs.Placebo over a period of 5 days
  Other Names: 0.1% Octenidine Mouthwash; OML
  Arms: Octenidine Mouthwash
Other: Placebo — Mouth rinsing of the oral cavity with Octenidinehydrochlorid vs.Placebo over a period of 5 days
  Arms: Placebo

SUMMARY:
The objective of the study is to demonstrate the superiority of 0.1% octenidine mouthwash (Octenidin Mundspüllösung, OML) to placebo (PLAC) in the inhibition of plaque formation. The study will consist of a 14-day screening period and a 5-day treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female subjects (aged 18 and older);
2. Subjects with a total mean gingival index1 (GI, Löe, 1967) ≤1.5 (0.0-1.5);
3. Subjects with at least 20 teeth (excluding wisdom teeth) with complete natural "Ramfjord-teeth" or their replacement teeth and 10 natural anterior teeth (excluding teeth provided with prosthetics such as crowns, dental bridges, veneers or large vestibular fillings such as large cervical or frontal teeth fillings; teeth with small interdental and orally oriented fillings are allowed);
4. Non-pigmented gingiva;
5. Signed informed consent.

Exclusion Criteria:

1. Subjects with severe systemic diseases (e.g. hepatitis, human immunodeficiency virus [HIV] infection, tuberculosis, acute cancer treatment);
2. Subjects who require endocarditis prophylaxis for dental examination and treatment;
3. Subjects with caries requiring treatment (e.g. caries with cavity) or other oral diseases (including gingival hyperplasia, diseases of the oral mucosa);
4. Subjects who have a history of chronic or aggressive periodontitis;
5. Subjects with current moderate or severe chronic or aggressive periodontitis (periodontal screening index [PSI] >2 in more than 2 sextants or PSI >3);
6. Subjects showing a GI score of 3 on at least one tooth;
7. Subjects who underwent oral surgery within 14 days prior to Screening;
8. Subjects who used antiseptic mouth rinse within 14 days prior to Screening;
9. Subjects wearing orthodontic appliances and removable dentures (Wire-retainers after orthodontic treatment are allowed);
10. Subjects treated with antibiotics less than 3 months prior to the baseline examination at Visit 1 and/or planning such treatment for the duration of the study;
11. Subjects treated with systemically acting corticosteroids or corticosteroids applied via the oral cavity (e.g. asthma sprays);
12. Subjects who suffer from xerostomia;
13. Subjects who have a known hypersensitivity or allergy to the test product and its ingredients or to medications that have a similar chemical structure;
14. Participation of the subject in another clinical study within the last 4 weeks before enrolment in and during this study;
15. Incapability of assessing essence and possible consequences of the study (e.g. alcoholism);
16. Pregnant or breastfeeding women;
17. Women with childbearing potential except those who fulfill one of the following criteria:

    1. Post-menopausal (12 months of natural amenorrhea or 6 months of amenorrhea with serum follicle-stimulating hormone [FSH] >40 U/ml);
    2. Postoperative (6 weeks after bilateral ovariectomy with or without hysterectomy);
    3. Continuous and correct application of a highly effective contraception method with a Pearl Index <1% (e.g. implants, depots, oral contraceptives, intrauterine device [IUD]);
    4. Sexual abstinence; whereas sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject;
    5. Confirmation of vasectomy of the sexual partner;
18. Evidence suggesting that the subject is not likely to follow the study protocol (e.g. lacking compliance).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Total mean PI (Plaque index according to Silness and Löe) after 5 days of treatment at Visit 2 | after 5 days of treatment
  The total mean PI is the sum of the individual scores divided by the number of investigated sites.

SECONDARY OUTCOMES:
Bacterial count reduction in saliva after a single administration of OML vs placebo | after 1 minute of rinsing
  Bacterial count in saliva will be assessed prior to the first administration of study medication and 1 min after the first administration
Change in total mean GI (Gingival Index according to Löe, 1967) from Visit 1 to Visit 2 | baseline and after 5 days of treatment
  The total mean GI is the sum of the individual scores divided by the number of investigated sites. The GI for each tooth is the sum of the 4 individual scores divided by 4.
Incidence and severity of AEs (adverse events) | 5 days
Incidence of SAEs (serious adverse events) | 15 days
Change in tooth discoloration index from Visit 1 to Visit 2 | baseline and after 5 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Jockel-Schneider, Dr.med.dent., Principal Investigator — Universitätsklinikum Würzburg, Poliklinik für Zahnerhaltung und Parodontologie
Locations (3):
- Universitätszahnklinik Wien, Fachbereich Zahnerhaltung und Parodontologie, Vienna, Austria
- Germany (2):
  - Poliklinik für Zahnerhaltung und Parodontologie des Universitätsklinikums Würzburg, Würzburg, Bavaria
  - Poliklinik für Zahnerhaltung und Parodontologie der Universitätsklinik Köln, Cologne, North Rhine-Westphalia